CLINICAL TRIAL: NCT04999527
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, PK and PD of DISC-0974 in Healthy Subjects Following Dose-Escalating Single Intravenous or Subcutaneous Administration
Brief Title: Study to Evaluate the Safety, Tolerability, PK and PD of DISC-0974 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Disc Medicine, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DISC-0974-101
Record Dates: First submitted 2021-07-20; First posted 2021-08-11 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteer: Single Ascending Dose of DISC-0974 (Experimental): Single Intravenous (IV) or Subcutaneous (SC) ascending dose in healthy volunteers
  Interventions: Drug: DISC-0974
- Healthy Volunteer: Single Ascending Dose of Placebo (Experimental): Single Intravenous (IV) or Subcutaneous (SC) ascending dose in healthy volunteers
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DISC-0974 — DISC-0974 is administered (IV infusion or Subcutaneous Injection) as a single dose
  Arms: Healthy Volunteer: Single Ascending Dose of DISC-0974
Drug: Placebo — Placebo is administered (IV infusion or Subcutaneous Injection) as a single dose
  Arms: Healthy Volunteer: Single Ascending Dose of Placebo

SUMMARY:
This Phase 1 study of DISC-0974 will assess the safety, tolerability, pharmacokinetics (PK) and Pharmacodynamics (PD) of DISC-0974 in adult healthy volunteers.

DETAILED DESCRIPTION:
Enrolled participants in this study will receive a single dose of DISC-0974 or a placebo. Samples will be collected to measure how DISC-0974 is processed by the body and how the body responds when exposed to DISC-0974. Participants will receive a single study drug dose on Day 1; and follow-up for 10 weeks (71 days). If an undetectable DISC-0974 blood concentration is observed, the duration of follow-up will be shortened to 7 days thereafter, as feasible.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (HV only) adults aged 18 to 65 years, inclusive at the time of consent.
* Body weight ≥50 kg and body mass index (BMI) between 18 and 33, inclusive, at Screening.
* Systolic blood pressure ≤140 mmHg and diastolic blood pressure ≤90 at Screening.
* No clinically significant abnormalities as determined by medical history, by results of physical examination, vital signs, ECG and lab tests at Screening.
* QTcF <450 msec at Screening.
* Estimated glomerular filtration rate >60 mL/min/1.73m2 based on the 4 parameter MDRD (Modification of Diet in Renal Disease) equation at Screening
* TSAT ≤30% at Screening, as determined in a fasting morning blood sample (06:00 to 11:00 hours).
* Hematologic parameters (red blood cell count [RBC], hemoglobin, hematocrit, platelet count, mean corpuscular volume, mean corpuscular hemoglobin concentration), serum iron, and TIBC within normal range and serum ferritin (within normal range and ≥30 ng/mL) at Screening.
* If a male with female sexual partner(s) of childbearing potential, must agree to use acceptable methods of birth control during the study and through the End of Study (EOS) visit
* If female, postmenopausal, as defined with at least 12 months natural, spontaneous amenorrhea, or at least 6 weeks following surgical menopause
* Able to understand and provide written informed consent and comply with protocol requirements

Exclusion Criteria:

* History of anemia or hematologic disorder within 1 year of Screening
* History of splenectomy
* Diagnosis or first-degree relative with a diagnosis of hemochromatosis
* History of diabetes, cardiovascular, hepatic, renal, or malabsorptive disease
* Vegan or iron-deficient diet within 3 months of Screening
* Blood transfusion within 1 year of Screening
* Whole blood donation within 6 months of Screening or plasma donation within 30 days of Screening.
* A history of alcohol or illicit drug use disorder within 3 years of Screening, as assessed by the Investigator
* Use of any tobacco- and/or nicotine-containing containing products, including e-cigarettes, vaping products, and nicotine replacement products, within 3 months of Screening
* Use of multivitamin or iron supplements within 30 days prior to Screening
* ALT or aspartate aminotransferase (AST) level above the normal range at Screening
* Positive urine pregnancy test at Screening or Baseline (Day -1).
* Positive serologic test for Hepatitis B surface antigen, Hepatitis C antibody, or human immunodeficiency virus (HIV) at Screening.
* Positive urine screen for drugs of abuse or alcohol test on admission to the study center
* Use of any systemic prescription medication within 14 days of Screening, non-iron containing dietary supplements, or non-prescription drugs within 7 days of dosing.
* History of a major surgical procedure within 60 days of Screening or planned surgical procedure within 90 days of dosing.
* A history or known allergic reaction to any investigational product excipients or history of anaphylaxis to any food or drug.
* History or presence or any illness that, in the opinion of the Investigator, would interfere with the ability to provide informed consent or comply with study instructions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 71 days of monitoring
Incidence of abnormal laboratory test results | Up to 71 days of monitoring
Incidence of treatment-emergent clinically abnormal electrocardiogram (ECG) | Up to 71 days of monitoring
Incidence of treatment-emergent clinically abnormal physical exam | Up to 71 days of monitoring

SECONDARY OUTCOMES:
Plasma maximum measured drug concentration (Cmax) | Up to 71 days of testing
Time of maximum concentration (Tmax) | Up to 71 days of testing
Area under the concentration-time curve (AUC) | Up to 71 days of testing
Plasma half-life (T½) | Up to 71 days of testing

CONTACTS AND LOCATIONS:
Overall Officials: William Savage, MD, PhD, Study Director — Disc Medicine
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

REFERENCES:
- [Derived] Novikov N, Buch A, Yang H, Andruk M, Liu G, Wu M, Howell H, MacDonald B, Savage W. First-in-Human Phase 1 Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of DISC-0974, an Anti-Hemojuvelin Antibody, in Healthy Participants. J Clin Pharmacol. 2024 Aug;64(8):953-962. doi: 10.1002/jcph.2432. Epub 2024 Mar 21. PMID 38515275
- See also: Related Info — https://www.discmedicine.com/